CLINICAL TRIAL: NCT02770352
Title: Assessment of Factors Surrounding Fistula Formation and Successful Repair at Bwaila Hospital, Lilongwe
Brief Title: Fistula Formation and Successful Repair
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 11-2345; CID 1116 (Other: UNC)
Record Dates: First submitted 2016-05-05; First posted 2016-05-12 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-02

CONDITIONS: Fistula; HIV
Keywords: retrospective chart review; prospective chart review; fistula formation and repair; database; demographics of women with fistulas; internationally accepted risks factors for fistula formation
MeSH Terms: conditions — Fistula

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this proposal is to create a database for obstetric fistula patients at Bwaila Hospital containing their demographics, obstetric history, fistula history, physical exam findings, intraoperative and postoperative results. Data collection will be prospective starting in 2011 upon institutional review board (IRB) approval to last a minimum of five years and will have a retrospective component tracing back to January 2010. Primary goals of data analysis will be to determine the risk factors for fistula formation, risk factors for poor surgical outcomes and long-term incontinence, social and economic impact of fistula repair, and the ability of various physical exam findings to predict likelihood of successful repair. It is expected that findings will lead to improved surgical management of obstetric fistulas both locally and internationally.

DETAILED DESCRIPTION:
This is a prospective and retrospective chart review of a cohort of women aged 12 years and above who present to Bwaila Hospital with obstetric fistulas. Variables from existing subject records tracing back to January 2010 will be input into the REDCap database and analyzed. Prospective data collection will begin alongside obstetric fistula repairs upon IRB approval and will last for a minimum of 5 years.

A few variables were selected from the database for sample size determination:

1. HIV prevalence In order to assess a statistically significant difference in HIV prevalence amongst fistula patients and the general population, with a projected prevalence of 25% in fistula patients and 15% in the general population based on prior studies, approximately 416 fistula patients would need to be enrolled in the study.
2. Risk factors for failure of repair-Goh classification Type 4 In order to assess a statistically significant difference in failure of repair for fistula patients classified based on the Goh classification as Type4 (approximately 30% failure rate based on prior studies) and all other fistula patients (15% failure rate reported for uncomplicated fistulas), approximately 200 patients would need to be enrolled in the study.

It is estimated that about 200 fistula patients will be enrolled into the database every year. The study is expected to last a minimum of 5 years, for a total enrollment of 1250 patients.

Current Procedures For more than a year, the Freedom to Fight Fistula Foundation (FFFF) has sponsored a fistula repair program at Bwaila that has consisted of visiting fistula surgeons coming for short periods of time to conduct repairs. Since September 2011, a full time fistula surgeon has been on site at Bwaila hospital.

Referral to the FFFF at Bwaila occurs primarily via word-of-mouth, as currently demand highly exceeds capacity. As of now, there is a waiting list of approximately 50 fistula patients. Occasionally, the foundation makes visits to health centers to give educational presentations on obstetric fistulas, and distributes flyers advertising its services in the local community. Once the presence of a regular surgeon is established, and the waiting list is diminished, the foundation anticipates increasing its advertising through newspaper and radio, and by making regular visits to community events and district health centers.

Bwaila Hospital is a hospital located in Lilongwe designated for women. It provides basic, regular obstetric and gynecologic services.

Data Collection and Bwaila Hospital

Retrospective Arm A chart review of existing subject records tracing back to January 2010 will be conducted, and input in the REDCap database to the extent that it is available and complete.

Prospective Arm Nurses will obtain informed consent from all patients admitted to Bwaila Hospital for obstetric fistula evaluation to participate in the research study.

They will then interview the patients with a clinical history form. The information collected with the form will be relevant to the care of the patient, and is part of routine care for obstetric fistula patients.

The form includes demographic data, sexual history, obstetric history, and medical history, and a depression screening and diagnostic tool.

After the interview the patient will receive standard of care with their obstetrics doctor for their fistulas (this is not part of the study): assessed for the presence of an obstetric fistula; discuss possible repair; have repair; recuperate; discharged; return for follow-up visits at one month and three months to assess how the patient is doing.

At these visits patient will have 5 minute study interviews discussing their ability to control their urination, and also how well they are getting by in their community, both financially and socially.

Additional data will be extracted directly from the patient chart as a secondary chart review for the study, and will include a review of physical exam findings, preoperative findings, intraoperative findings, postoperative results and follow-up findings at the one-month and three-month review dates.

This data will be transferred from the patient charts to REDCap. All information collected will be de-identified.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 12 years and above
* Present to Bwaila Hospital with obstetric fistula
* Allow retrospective chart review
* Willing to provide consent

Exclusion Criteria:

* Not allow retrospective chart review

Ages: 12 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants are women admitted to Bwaila Hospital for repair of obstetric fistulas.
Sampling Method: Non-Probability Sample
Enrollment: 1817 (Actual)
Dates: Start 2012-10; Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

PRIMARY OUTCOMES:
Successful obstetric fistula repair | 3-months after obstetric fistula repair
  Successful obstetric fistula repair is defined by having a negative dye test (no leakage of dye into the vagina after dye is infused into the bladder). Factors associated with successful obstetric fistula repair will be evaluated.

SECONDARY OUTCOMES:
Rates of depression among women undergoing obstetric fistula repair and associated factors | 3-months after obstetric fistula repair
  Participants will complete the patient health questionnaire (PHQ)-9, a standardized tool to diagnose depression before and after obstetric fistula repair. Factors associated with post-operative depression will be explored such as HIV, number of living children, and marital status.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Tang, MD, MSCR, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Project, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: No